CLINICAL TRIAL: NCT06492668
Title: Risk of Exposure and Prevention of Ticks and Tick-borne Diseases Among Foresters in Alsace (France)
Brief Title: Risk of Exposure and Prevention of Ticks and Tick-borne Diseases Among Foresters in Alsace
Acronym: PREFORTIC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9309
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Lyme Borreliosis
Keywords: Tick-Borne Diseases; Lyme borreliosis; Febrile syndromes; Ixodes ricinus tick
MeSH Terms: conditions — Lyme Disease; Tick-Borne Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ticks are blood-sucking arthropods that feed on vertebrate hosts. Although wild and domestic animals are the primary source of tick blood meals, humans can be an accidental host. During a blood meal, a microorganism can be transmitted to the host who can develop a disease. All infectious diseases transmitted by ticks are referred to as tick-borne diseases (TBDs). They are the most prevalent vector-borne diseases in the Northern Hemisphere. Among these diseases, Lyme borreliosis is the most common.

In Europe, Lyme borreliosis does not cause high fevers (> 38°C). Therefore, when a patient presents with a high fever with the notion of exposure to ticks, another etiology must be suspected. Anaplasma phagocytophilum and the tick-borne encephalitis virus are classically described as causing febrile syndromes.

In France, ticks and tick-borne diseases are increasing, particularly those associated with the Ixodes ricinus tick. This tick is mainly present in forest ecosystems with a peak of activity in May. Foresters represent a population with biting ticks and tick-borne diseases, notably Lyme borreliosis.

ELIGIBILITY:
Inclusion Criteria:

* Major forester (≥18 years old)
* Male or female gender
* ONF (National Forestry Office) staff
* Regularly exposed to ticks in Alsace (exclusively)
* Practicing regular forestry activities in a group
* Agreeing to participate in the study.

Exclusion criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major forester (≥18 years old), ONF (National Forestry Office) staff regularly exposed to ticks in Alsace.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07-08 (Estimated)

PRIMARY OUTCOMES:
Number of ticks found on clothing during activities in forest ecosystems, and if tick bites, their number. | 1 year
  This study is carried out on foresters in the Alsacce region over a period of one year.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre National de Référence Borrelia - CHU de Strasbourg - France, Strasbourg, Les Hôpitaux Universitaires de Strasbourg, France